CLINICAL TRIAL: NCT02181894
Title: Identifying the Most Accurate Method for Predicting the Safe Depth of Orally Placed Neonatal Endotracheal Tubes.
Brief Title: Identifying the Most Accurate Method for Predicting the Safe Depth of Orally Placed Neonatal Endotracheal Tubes (ETT).
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 14-1117; UL1TR001082 (NIH)
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Infant Showing No Response to Resuscitation; Ventilator Adverse Event; Apparent Life Threatening Event in Newborn and Infant
Keywords: Infant; Newborn; Neonate; Intubation; Neonatal resuscitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Orally intubated infants: Subjects will be <72 hours of age and orally intubated. Following consent, four measures will be reported (i.e. body weight, nasal to tragus length, suprasternal notch to xyphoid process and shoulder to elbow length). Measures will be compared against a chest x-ray and placement of ETT at the subjects lip to identify the most accurate method to place endotracheal tubes in the newborn.

SUMMARY:
Placing artificial airways in infants is often performed under emergent life-saving conditions, which necessitates a procedure that is both accurate and efficient. Intubations of the newborn are often necessary before an accurate weight can be reported and estimations are often inaccurate. The current national standard uses body weight to predict the appropriate tube depth yet this approach tends to place the tube too deep for the smallest and most vulnerable neonate; and placement accuracy of any size infant is only 50-70%. The consequence of malpositioned ETTs resulting from poor oxygenation, lung hyperinflation, pneumothoraces and death has been suggested to cost $20 to $54 million annually.

The morbidity and the financial impact suggest an optimal and accurate approach to place ETT in neonates has not been identified. Other methods to estimate the proper depth of the orotracheal tube have shown promise yet no comparison studies have been performed. Identifying the most accurate method to safely place neonatal orotracheal tubes will improve placement precision and reduce adverse events and their associated costs.

Hypothesis

Compared to weight, sternal to xyphoid length and shoulder to elbow length, the nasal to tragus length will become the most accurate method for predicting the safe depth of orally placed neonatal endotracheal tubes.

ELIGIBILITY:
Inclusion Criteria:

* Infants orally intubated and admitted into the Neonatal Intensive Care Unit.

Exclusion Criteria:

* Previous intubation
* Hydrops fetalis
* Thoracic congenital anomalies
* Facial abnormalities
* Naso-tracheal intubation

Ages: 1 Minute to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants <72 hours of age and orally intubated
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2014-11; Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
The differences between 4 measurement methods in placing a neonatal ETT between the lower border of T1 and upper margin of T3 on chest radiograph. | Up to 3 years

SECONDARY OUTCOMES:
The differences in head position in placing a neonatal ETT between the lower border of T1 and upper margin of T3 on chest radiograph. | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Moran, DNP APRN NNP-BC FFNMRCSI, Principal Investigator — Children's Hospital Colorado
Locations (5):
- United States (3):
  - Kaiser Permanente, Los Angeles Medical Center, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
- Ireland (2):
  - The Coombe Women & Infants University Hospital, Dublin
  - The Rotunda Hospital, Dublin